CLINICAL TRIAL: NCT01265589
Title: Intratracheal Vitamin A Administration With Surfactant for Newborn Respiratory Distress Syndrome
Acronym: RDS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Third Military Medical University (Other)
Responsible Party: Yuan Shi and Heqiang Sun, Daping Hospital, Third Military Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2011001
Record Dates: First submitted 2010-12-03; First posted 2010-12-23 (Estimated); Last update posted 2011-07-26 (Estimated); Status verified 2010-11

CONDITIONS: RDS; Infant, Newborn; Vitamin A; Surfactant
Keywords: RDS; Infant, newborn; Vitamin A; Surfactant
MeSH Terms: interventions — Surface-Active Agents

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- I=surfactant (Placebo Comparator): Intratracheal Surfactant Administration without Vitamin A for Newborn Respiratory Distress Syndrome
  Interventions: Drug: surfactant
- II=surfactant+vitamin A (Experimental): Intratracheal Surfactant Administration with Vitamin A for Newborn Respiratory Distress Syndrome
  Interventions: Drug: surfactant+vitamin A

INTERVENTIONS:
Drug: surfactant — Intratracheal Surfactant Administration without Vitamin A for Newborn Respiratory Distress Syndrome
  Arms: I=surfactant
Drug: surfactant+vitamin A — Intratracheal Surfactant Administration with Vitamin A for Newborn Respiratory Distress Syndrome
  Arms: II=surfactant+vitamin A

SUMMARY:
To research the effect of vitamin A to newborn respiratory distress syndrome by intratracheal administration with surfactant.

DETAILED DESCRIPTION:
Chronic lung disease (CLD) of prematurity is the major cause of long-term disability of extremely LBW (ELBW) premature infants, and it is the most cost consumptive disease in Neonatal Intensive Care Unit graduates. Vitamin A plays an important role in the development of premature lung. Nevertheless, premature infants are prone to vitamin A deficiency. Oral supplementation of vitamin A does not alter the incidence of CLD in ELBW infants. Intramuscular administration of vitamin A reduced the incidence of CLD. The treatment is considered painful and this way is not routinely practiced. Vitamin A is systemically bioavailable after intratracheal administration with surfactant in an animal model of newborn respiratory distress.

ELIGIBILITY:
Inclusion Criteria:

* 1.Newborn infants with birth weight >500 gm.
* 2.Gestational age >24 completed weeks.
* 3.Intention to manage the infant with non-invasive respiratory support (i.e. no endotracheal tube), where either: 1) the infant is within the first 7 days of life and has never been intubated or has received less than 24 hours of total cumulative intubated respiratory support; 2)the infant is within the first 28 days of life, has been managed with intubated respiratory support for 24 hours or more and is a candidate for extubation followed by non-invasive respiratory support.
* 4.No known lethal congenital anomaly or genetic syndromes.
* 5.Signed parental informed consent

Exclusion Criteria:

* 1.Considered non-viable by clinician (decision not to administer effective therapies)
* 2.Life-threatening congenital abnormalities including congenital heart disease (excluding patent ductus arteriosis)
* 3.Infants known to require surgical treatment
* 4.Abnormalities of the upper and lower airways
* 5.Neuromuscular disorders
* 6.Infants who are >28 days old and continue to require mechanical ventilation with an endotracheal tube

Max Age: 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2012-01; Primary Completion 2012-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Intratracheal Vitamin A Administration with Surfactant for Newborn Respiratory Distress Syndrome | 1 year
  get the date of infants' reflects with Intratracheal Vitamin A Administration

SECONDARY OUTCOMES:
Overall clinical outcomes at Newborn Infants With Respiratory Distress Syndrome | 13 months
  analysis the date and drow a conclusion

CONTACTS AND LOCATIONS:
Overall Officials: Yuan Shi, MD, Study Director — Department of Pediatrics, Daping Hospital, Third Military Medical University
Locations (1):
- Deaprtment of Pediatrics, Daping Hospital, Third Military Medical University, Chongqing, Chongqing Municipality, China